CLINICAL TRIAL: NCT01872312
Title: The Humanatarian Use of the Spiration IBV® Valve System and Spiration Airway Sizing Kit for Use in Patients at The Ohio State University Medical Center.
Brief Title: Spiration IBV® Valve System and Spiration Airway Sizing Kit
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not sure. PI is no longer at OSU.
Sponsor: Ohio State University (Other)
Collaborators: Olympus Corporation of the Americas (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012H0033
Record Dates: First submitted 2013-04-10; First posted 2013-06-07 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Management of BPF (Bronchopleural Fistulae)
Keywords: BPF(Bronchopleural fistulae)
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Other): Loading IBV® Valve System
  Interventions: Device: treatment with valves (The Spiration® IBV Valve System)

INTERVENTIONS:
Device: treatment with valves (The Spiration® IBV Valve System) — treat BPF
  Other Names: spiration valve; IBV Valve System

SUMMARY:
This procedure allows patients to use the Humanitarian Use Device, IBV® Valve System.

DETAILED DESCRIPTION:
IBV® Valve System The Spiration® IBV Valve System is a device to control prolonged air leaks of the lung, or significant air leaks that are likely to become prolonged air leaks following lobectomy, segmentectomy, or lung volume reduction surgery (LVRS). An air leak present on postoperative day 7 is considered prolonged unless present only during forced exhalation or cough. An air leak present on day 5 should be considered for treatment if it is: 1) continuous, 2) present during normal inhalation phase of inspiration, or 3) present upon normal expiration and accompanied by subcutaneous emphysema or respiratory compromise. IBV Valve System use is limited to 6 weeks per prolonged air leak.

ELIGIBILITY:
Inclusion Criteria:

* Unresolved BPF
* Not candidate for surgical repair

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03-25 (Actual); Primary Completion 2014-02-14 (Actual); Study Completion 2014-02-14 (Actual)

PRIMARY OUTCOMES:
resolution of BPF (Bronchopleural Fistulae) | 6 weeks
  expected resolution of BPF (Bronchopleural Fistulae) in three weeks
resolutin of BPF | 6 weeks
  anticipated the with the use of valves the BPF would improve and the valves can be removed in 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: shaheen Islam, MD, Principal Investigator — Ohio State University
Locations (1):
- OSUMC, Columbus, Ohio, United States